CLINICAL TRIAL: NCT04584411
Title: Patterns of Arrhythmias and Conduction Block in COVID-19 Patients and Its Relation to Myocardial Injury Detected by Cardiac Magnetic Resonance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Rahim Hassaan, resident, Assiut University
Other Study IDs: arrhythmias in COVID-19
Record Dates: First submitted 2020-09-09; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic resonance imaging — The following basic sequences will be conducted:
  * Cine imaging using SSFP sequence for cardiac structure and function.
  * Tissue characterization imaging, T1 and T2.
  * Myocardial perfusion imaging.
  * Late gadolinium enhancement.
  Diagnosis of myocarditis will be based on the modified Lake Louise criteria:
  T2-weighted: any of the following standard T2 sequences: regional high signal standard T2 sequences: global signal intensity ratio (myocardium/skeletal muscle) ≥2 T2 mapping: increased T2 relaxation times T1-weighted: any of the following late enhancement imaging: non-ischemic (subepicardial or mid myocardial) late enhancement native T1 mapping: increased T1 relaxation times or extracellular volume supportive criteria: signs of pericarditis: effusion or pericardial late enhancement regional or global wall motion abnormalities[5]

SUMMARY:
Detection of the incidence and types of arrhythmia and conduction block in COVID - 19 patients Detection and description of CMR patterns of myocardial injury in COVID-19 patients with arrhythmias.

DETAILED DESCRIPTION:
COVID-19 has been declared a global pandemic by the World Health Organization and is responsible for hundreds of thousands of deaths worldwide.

Early reports from China suggested an overall cardiac arrhythmia incidence of 17% in patients hospitalized for COVID-19. A higher arrhythmia rate (44%) was observed in patients with COVID-19 admitted to the intensive care unit (ICU). However, details of the type and burden of arrhythmias in this population have not been elucidated.

Myocardial injury is common in patients with COVID-19, accounting for 7%-23% of reported cases in Wuhan, China. Among COVID-related myocardial injury, etiologies vary and can include myocarditis, myocardial infarction, sepsis-related myocardial injury, and/or stress induced cardiomyopathy. Myocardial injury is associated with high risk of developing all types of arrhythmia including atrial fibrillation, supraventricular tachycardia, ventricular tachycardia, ventricular fibrillation, and variable degrees of heart block. Sudden cardiac death was also reported.

The pathophysiology of COVID-19-related myocarditis is a combination of direct viral injury and cardiac damage due to the host's immune response. Although the pathophysiology of arrhythmias is still speculative, clinicians should provide prompt monitoring and treatment. The long term impact of COVID-19 myocarditis remains unknown

Meanwhile, cardiac magnetic resonance (CMR) imaging is an integral test in the diagnosis of myocardial injury. It can safely be used as a first-line diagnostic tool in the workup of myocardial injury associated with COVID-19.

Investigators believe that proper diagnosis and management of COVID 19 related arrhythmias and their etiology can lead to both in-hospital and long term reduction of morbidity and mortality of this dangerous presentation of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. COVID 19 suspected patients presented by chest pain, dyspnea, chest discomfort &/or palpitations
2. ECG changes (LBBB, PVCs, ventricular tachycardia, AF, atrial flutter, ST-T changes, and conduction defects).
3. Increased inflammatory markers and / or Tropnin-I.

Exclusion Criteria:

1. COVID 19 patients without ECG changes.
2. Patients known to have the same pattern of arrhythmia or conduction system defects before Covid-19 infection.
3. Patients contraindicated for CMR.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 50 confirmed COVID-19 patients admitted to Assiut University Heart Centre and critical care unit, internal medicine department within the next 6 months complaining of arrhythmias and heart block. These patients will be followed-up for a period of 6 months after discharge.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the incidence of arrhythmia and conduction block in COVID-19 patients using Holter | baseline

SECONDARY OUTCOMES:
Detection of myocardial injury in COVID-19 patients using CMR. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Fouad, Doctorate, Principal Investigator — Assiut University; Alaa A El-Moniem, Doctorate, Principal Investigator — Assiut University; Mohamed A.H Abdelhafez, Doctorate, Principal Investigator — Assiut University; Shimaa S Khider, Doctorate, Principal Investigator — Assiut University; Ahmed AR Hassaan, bachelor, Principal Investigator — Assiut University; Maram M Shafiq, student, Principal Investigator — Assiut University

REFERENCES:
- [Background] Pirzada A, Mokhtar AT, Moeller AD. COVID-19 and Myocarditis: What Do We Know So Far? CJC Open. 2020 May 28;2(4):278-285. doi: 10.1016/j.cjco.2020.05.005. eCollection 2020 Jul. PMID 32691024
- [Background] Bhatla A, Mayer MM, Adusumalli S, Hyman MC, Oh E, Tierney A, Moss J, Chahal AA, Anesi G, Denduluri S, Domenico CM, Arkles J, Abella BS, Bullinga JR, Callans DJ, Dixit S, Epstein AE, Frankel DS, Garcia FC, Kumareswaram R, Nazarian S, Riley MP, Santangeli P, Schaller RD, Supple GE, Lin D, Marchlinski F, Deo R. COVID-19 and cardiac arrhythmias. Heart Rhythm. 2020 Sep;17(9):1439-1444. doi: 10.1016/j.hrthm.2020.06.016. Epub 2020 Jun 22. PMID 32585191
- [Background] Shirazi S, Mami S, Mohtadi N, Ghaysouri A, Tavan H, Nazari A, Kokhazadeh T, Mollazadeh R. Sudden cardiac death in COVID-19 patients, a report of three cases. Future Cardiol. 2021 Jan;17(1):113-118. doi: 10.2217/fca-2020-0082. Epub 2020 Jul 3. PMID 32615807
- [Background] B. Siripanthong et al., "Since January 2020 Elsevier has created a COVID-19 resource centre with free information in English and Mandarin on the novel coronavirus COVID- company ' s public news and information website . Elsevier hereby grants permission to make all its COVID-19-r," no. January, 2020.
- [Background] Ferreira VM, Schulz-Menger J, Holmvang G, Kramer CM, Carbone I, Sechtem U, Kindermann I, Gutberlet M, Cooper LT, Liu P, Friedrich MG. Cardiovascular Magnetic Resonance in Nonischemic Myocardial Inflammation: Expert Recommendations. J Am Coll Cardiol. 2018 Dec 18;72(24):3158-3176. doi: 10.1016/j.jacc.2018.09.072. PMID 30545455